CLINICAL TRIAL: NCT06205056
Title: Phase I, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of an Ad26.Mos4.HIV and CH505 TF chTrimer (Env) Combination to Mimic Acute HIV Viral Replication Kinetics in Healthy Adults
Brief Title: Evaluation of Safety and Immunogenicity of Ad26.Mos4.HIV and CH505 TF chTrimer Combination in Healthy Adults
Acronym: RV591
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Janssen Vaccines & Prevention B.V. (Industry); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other); Duke University (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Makerere University Walter Reed Project (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: S-22-03; W81XWH-18-2-0040 (Other Grant/Funding Number: DAIDS/NIAID/NIH)
Record Dates: First submitted 2023-10-10; First posted 2024-01-12 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ad26.Mos4.HIV and CH505 TF chTrimer + ALFQ [Arm 1a] (Experimental): Arm 1a [Co-administration]: Dose consistent injections (5x10^10 vp/0.5 mL) of Ad26.Mos4.HIV in a 0.5 mL injection volume and dose consistent injections of CH505 TF chTrimer (300 µg)+ALFQ (200 µg MPLA/100 µg QS-21) in a 1.1 mL injection volume on Study Days 1 and 57, followed by a dose-consistent injection of CH505 TF chTrimer (300 µg)+ALFQ (200 µg MPLA/100 µg QS 21) in a 1.1 mL injection volume on Study Day 169 (11 participants) OR a 0.5 mL injection and a 1.1 mL injection of Placebo on Study Days 1 and 57, followed by a 1.1 mL injection of Placebo on Study Day 169 (3 participants)
  Interventions: Biological: Ad26.Mos4.HIV in CH505 TF chTrimer + ALFQ [Arm 1a]; Biological: CH505 TF chTrimer + ALFQ [Arm 1a]; Biological: Placebo [Arm 1a]
- CH505 TF chTrimer + ALFQ [Arm 1b] (Experimental): Arm 1b [Trimer Bolus Administration]: Dose consistent injections of CH505 TF chTrimer (300 µg)+ALFQ (200 µg MPLA/100 µg QS-21) in a 1.1 mL injection volume on Study Days 1, 57, and 169 (20 participants) OR a 1.1 mL injection of Placebo on Study Days 1, 57, and 169 (5 participants)
  Interventions: Biological: CH505 TF chTrimer + ALFQ [Arm 1b]; Biological: Placebo [Arm 1b]
- Ad26.Mos4.HIV and CH505 TF chTrimer + ALFQ [Arm 2a] (Experimental): Arm 2a [Rapidvax]: A lower dose of Ad26.Mos4.HIV (2.5x10^10 vp/0.25mL) in a 0.25mL injection volume (InjV) + lower dose of CH505 TF chTrimer (30 µg)+ALFQ (50µg MPLA/25µg QS-21) in a 0.5mL InjV [Study Day (SD) 1]; followed by rapid, dose escalating injections of CH505 TF chTrimer (100µg, 150µg, and 300µg)+ALFQ (50µg MPLA/25µg QS-21) on SD's 4, 8 (0.5mL InjV), and 15 (0.9mL InjV); followed by injections of Ad26.Mos4.HIV (5x10^10 vp/0.5mL) in a 0.5mL InjV + CH505 TF chTrimer (300µg)+ALFQ (200µg MPLA/100µg QS 21) in a 1.1mL InjV on SD 57; followed by an injection of CH505 TF chTrimer (300µg)+ALFQ (200µg MPLA/100µg QS 21) in a 1.1mL InjV on SD 169 (11 participants) OR a 0.25mL injection and a 0.5mL injection of Placebo [P] on SD 1; followed by 0.5mL, 0.5mL, and 0.9 mL injections of [P] on SD's 4, 8, and 15, respectively; followed by a 0.5mL injection + 1.1mL injection of [P] on SD 57; followed by a 1.1mL injection of [P] on SD 169 (3 participants)
  Interventions: Biological: Ad26.Mos4.HIV in CH505 TF chTrimer +ALFQ [Arm 2a]; Biological: CH505 TF chTrimer +ALFQ [Arm 2a]; Biological: Placebo [Arm 2a]
- CH505 TF chTrimer + ALFQ [Arm 2b] (Experimental): Arm 2b [Trimer Rapidvax]: A lower dose of CH505 TF chTrimer (30 µg)+ALFQ (50 µg MPLA/25 µg QS 21) in a 0.5 mL injection volume on Study Day 1; followed by rapid, dose escalating injections of CH505 TF chTrimer (100 µg, 150 µg, and 300 µg)+ALFQ (50 µg MPLA/ 25 µg QS-21) on Study Days 4 (0.5 mL injection volume), 8 (0.5 mL injection volume), and 15 (0.9 mL injection volume); followed by injections of CH505 TF chTrimer (300 µg)+ALFQ (200 µg MPLA/100 µg QS 21) in a 1.1 mL injection volume on Study Days 57 and 169 (20 participants); OR a 0.5 mL injection of Placebo on Study Days 1, 4, and 8; followed by a 0.9 mL injection of Placebo on Study Day 15; followed by a 1.1 mL injection of Placebo on Study Days 57 and 169 (5 participants)
  Interventions: Biological: CH505 TF chTrimer + ALFQ [Arm 2b]; Biological: Placebo [Arm 2b]

INTERVENTIONS:
Biological: Ad26.Mos4.HIV in CH505 TF chTrimer + ALFQ [Arm 1a] — Participants in Arm 1a will receive dose consistent injections (5x10^10 vp/0.5 mL) of Ad26.Mos4.HIV in a 0.5 mL injection volume and dose consistent injections of CH505 TF chTrimer (300 µg)+ALFQ (200 µg MPLA/100 µg QS-21) in a 1.1 mL injection volume on Study Days 1 and 57
  Arms: Ad26.Mos4.HIV and CH505 TF chTrimer + ALFQ [Arm 1a]
Biological: CH505 TF chTrimer + ALFQ [Arm 1a] — Participants in Arm 1a will receive a dose-consistent injection of CH505 TF chTrimer (300 µg)+ALFQ (200 µg MPLA/100 µg QS 21) in a 1.1 mL injection volume on Study Day 169.
  Arms: Ad26.Mos4.HIV and CH505 TF chTrimer + ALFQ [Arm 1a]
Biological: Placebo [Arm 1a] — Participants in Arm 1a will receive dose-consistent 0.5 mL injection and a 1.1 mL injection of Placebo on Study Days 1 and 57, followed by a 1.1 mL injection of Placebo on Study Day 169.
  Arms: Ad26.Mos4.HIV and CH505 TF chTrimer + ALFQ [Arm 1a]
Biological: Ad26.Mos4.HIV in CH505 TF chTrimer +ALFQ [Arm 2a] — Participants in Arm 2a will receive a lower dose of Ad26.Mos4.HIV (2.5x10^10 vp/0.25 mL) in a 0.25 mL injection volume and a lower dose of CH505 TF chTrimer (30 µg)+ALFQ (50 µg MPLA/25 µg QS-21) in a 0.5 mL injection volume on Study Day 1.
  Participants in Arm 2a will receive an injection Ad26.Mos4.HIV (5x10^10 vp/0.5 mL) in a 0.5 mL injection volume and CH505 TF chTrimer (300 µg)+ALFQ (200 µg MPLA/100 µg QS 21) in a 1.1 mL injection volume on Study Day 57.
  Arms: Ad26.Mos4.HIV and CH505 TF chTrimer + ALFQ [Arm 2a]
Biological: CH505 TF chTrimer +ALFQ [Arm 2a] — Participants in Arm 2a will receive a rapid, dose escalating injections of CH505 TF chTrimer (100 µg, 150 µg, and 300 µg)+ALFQ (50 µg MPLA/ 25 µg QS-21) on Study Days 4 (0.5 mL injection volume), 8 (0.5 mL injection volume), and 15 (0.9 mL injection volume).
  Participants in Arm 2a will receive a injection of CH505 TF chTrimer (300 µg)+ALFQ (200 µg MPLA/100 µg QS 21) in a 1.1 mL injection volume on Study Day 169.
  Arms: Ad26.Mos4.HIV and CH505 TF chTrimer + ALFQ [Arm 2a]
Biological: Placebo [Arm 2a] — Participants in Arm 2a will receive a 0.25 mL injection and a 0.5 mL injection of Placebo on Study Day 1; followed by 0.5 mL, 0.5 mL, and 0.9 mL injections of Placebo on Study Days 4, 8, and 15, respectively; followed by a 0.5 mL injection and a 1.1 mL injection of Placebo on Study Day 57; followed by a 1.1 mL injection of Placebo on Study Day 169.
  Arms: Ad26.Mos4.HIV and CH505 TF chTrimer + ALFQ [Arm 2a]
Biological: CH505 TF chTrimer + ALFQ [Arm 1b] — Participants in Arm 1b will receive dose consistent injections of CH505 TF chTrimer (300 µg)+ALFQ (200 µg MPLA/100 µg QS-21) in a 1.1 mL injection volume on Study Days 1, 57, and 169.
  Arms: CH505 TF chTrimer + ALFQ [Arm 1b]
Biological: Placebo [Arm 1b] — Participants in Arm 1b will receive a 1.1 mL injection of Placebo on Study Days 1, 57, and 169.
  Arms: CH505 TF chTrimer + ALFQ [Arm 1b]
Biological: CH505 TF chTrimer + ALFQ [Arm 2b] — Participants in Arm 2b will receive a lower dose of CH505 TF chTrimer (30 µg)+ALFQ (50 µg MPLA/25 µg QS 21) in a 0.5 mL injection volume on Study Day 1.
  Participants in Arm 2b will receive a rapid, dose escalating injections of CH505 TF chTrimer (100 µg, 150 µg, and 300 µg)+ALFQ (50 µg MPLA/ 25 µg QS-21) on Study Days 4 (0.5 mL injection volume), 8 (0.5 mL injection volume), and 15 (0.9 mL injection volume).
  Participants in Arm 2b will receive a injections of CH505 TF chTrimer (300 µg)+ALFQ (200 µg MPLA/100 µg QS 21) in a 1.1 mL injection volume on Study Days 57 and 169.
  Arms: CH505 TF chTrimer + ALFQ [Arm 2b]
Biological: Placebo [Arm 2b] — Participants in Arm 2b will receive a 0.5 mL injection of Placebo on Study Days 1, 4, and 8; followed by a 0.9 mL injection of Placebo on Study Day 15; followed by a 1.1 mL injection of Placebo on Study Days 57 and 169.
  Arms: CH505 TF chTrimer + ALFQ [Arm 2b]

SUMMARY:
This is a Phase I, randomized, double-blind, placebo-controlled clinical study to define the safety and immunogenicity resulting from a rapid dose-escalating vaccination schedule as compared to that of a co-administered, dose-consistent vaccination schedule. Participants randomized to receive vaccines will get either dose-consistent injections of CH505 TF chTrimer+ALFQ co-administered with Ad26.Mos4.HIV or rapid, dose-escalating injections of CH505 TF chTrimer+ALFQ with an Ad26.Mos4.HIV prime, followed by dose-consistent injection of CH505 TF chTrimer+ALFQ co-administered with Ad26.Mos4.HIV

DETAILED DESCRIPTION:
This study is exploratory and will be a randomized, placebo-controlled, double-blind trial. A total of 78 healthy male and female participants, aged 18 to 50 years, who are at low risk for Human Immunodeficiency Virus (HIV) acquisition will be enrolled and randomized across four Arms (1a, 2a, 1b, and 2b). Enrollment will be completed in two parts, dubbed Part A and Part B. In Part A, up to 28 participants will be randomized across Arms 1a and 2a, with up to 14 participants per Arm. Within these Arms, participants will be randomized 11:3 to active vaccine versus placebo (normal saline) and followed for up to 18 months. In Part B, participants will be randomized across Arms 1b and 2b, with 25 individuals per Arm. Within these Arms, participants will be randomized 4:1 to active study vaccine versus placebo (normal saline) and followed for up to 18 months. All products will be administered by intramuscular (IM) injection into the same quadriceps muscle at each product administration visit.

Participants randomized to receive active study vaccines in Arm 1a will receive dose-consistent injections of Ad26.Mos4.HIV (5x1010 viral particles [vp]/0.5 mL) and CH505 TF chTrimer (300 µg)+ALFQ (200 µg MPLA/100 µg QS 21) co administered on Study Days 1 and 57, followed by a dose-consistent injection of CH505 TF chTrimer (300 µg)+ALFQ (200 µg MPLA/100 µg QS 21) on Day 169.

Participants randomized to receive active study vaccines in Arm 2a will receive a lower dose of Ad26.Mos4.HIV (2.5x1010 vp/0.25 mL) and CH505 TF chTrimer (30 µg)+ALFQ (50 µg MPLA/25 µg QS 21) on Study Day 1, followed by rapid dose escalating injections of CH505 TF chTrimer (100 µg, 150 µg, and 300 µg)+ALFQ (50 µg MPLA/25 µg QS 21) through Study Day 15, followed by injections of Ad26.Mos4.HIV (5x1010 vp/0.5 mL) and CH505 TF chTrimer (300 µg)+ALFQ (200 µg MPLA/100 µg QS 21) on Study Day 57, followed by an injection of CH505 TF chTrimer (300 µg)+ALFQ (200 µg MPLA/100 µg QS 21) on Study Day 169.

Participants randomized to receive active study vaccines in Arm 1b will have a similar dosing regimen as participants in Arm 1a but without Ad26.Mos4.HIV on Study Days 1 and 57.

Participants randomized to receive active study vaccines in Arm 2b will have a similar dosing regimen as participants in Arm 2a but without Ad26.Mos4.HIV on Study Days 1 and 57.

Enrollment into Arms 1a and 2a will be concurrent. Sentinel groups, comprised of the first eight participants enrolled across Arms 1a and 2a (4 participants per Arm; 3:1 active vaccine to placebo in each Arm), will be included to facilitate an assessment of the safety of the combination of products and vaccination regimens. For each sentinel group, the Safety Monitoring Committee (SMC) will review safety data, covering a period of 7 days post-injection, to determine if it is safe to continue enrollment in that Arm. For participants in Arm 1a, this includes safety data from immediately after the first study injection through Day 8. For participants in Arm 2a, this includes safety data from immediately after the first injection through Day 22 (i.e., through 7 days post-Day 15 injection). While Arm 1a and Arm 2a sentinel safety reviews can occur separately, safety data from both Arms will be considered. For Arms 1a and 2a, the remaining 20 participants (10 per Arm) will be enrolled at a rate of up to 3 participants per week (up to 2 in the first week after re-initiation of enrollment) only after the SMC confirms that it is safe to continue, and the Sponsor gives their approval to proceed.

Enrollment in Part B (i.e., Arms 1b and 2b) will be initiated after enrollment in Part A (i.e., Arms 1a and 2a) has concluded, the SMC confirms that it is safe to continue after reviewing 7- or 21-days of post injection safety data from all Part A participants, and the Sponsor gives their approval to proceed. Part B enrollment will be similar to that in Part A, including concurrent enrollment into Arms 1b and 2b; the inclusion of sentinel groups, comprised of the first eight participants enrolled across Arms 1b and 2b (4 participants per Arm; 3:1 active vaccine to placebo in each Arm); and SMC review once 7- or 21-days of post-injection safety data is available from Arm 1b and 2b sentinel groups, respectively. Enrollment of the remaining 42 participants (21 per Arm) will occur only after the SMC confirms that it is safe to continue, and the Sponsor gives their approval to proceed.

Enrollment in Part B will be restricted to a rate of up to 3 participants per week; however, the rate of enrollment may increase if, based on available safety data the risk to participants will not be negatively impacted, and only if approved by the Sponsor.

Inguinal lymph node biopsies will be performed on Study Day 71 in a subset of participants from all four study Arms who provide consent for the optional procedure.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for participation:

1. Male or female, aged 18 to 50 years, inclusive, at the time of enrollment
2. Willing and able to read, sign, and date the informed consent form
3. Demonstrates an understanding of the study with a passing score (90% or greater) on the TOU by the third attempt, before study-related procedures are performed
4. Willing and able to comply with study requirements and be available to attend visits for the duration of study participation
5. Must have the means to be contacted by telephone for the duration of study participation
6. Willing to have photo or fingerprint taken for identification purposes
7. At low risk for HIV acquisition per investigator assessment
8. Agrees to refrain from donating blood or plasma outside of this study for at least the duration of study participation
9. Healthy based on the physician investigator's clinical judgment after review of past medical history, medication use, vital signs, and an abbreviated physical examination

   Note: Good health is defined by the absence of any medical condition described in the exclusion criteria in a participant with a normal abbreviated physical exam and vital signs. If the participant has a preexisting chronic condition not listed in the exclusion criteria, the condition cannot meet any of the following criteria:
   1. first diagnosed within the 12 weeks prior to screening; or
   2. worsening in terms of clinical outcome in the 24 weeks prior to screening; or
   3. involves the need for medication that may pose a risk to the participant's safety or impede assessment of adverse events or immunogenicity if they participate in the study.

   Note: Vital signs must be normal by Adverse Event Grading Scales, local normal ranges, or determined to be a normal variant by the physician investigator.

   Note: An abbreviated physical exam differs from a complete exam in that it does not include a genitourinary and rectal exam.
10. Laboratory criteria within 45 days prior to enrollment:

    1. Hemoglobin ≥11.0 g/dL for females; ≥12.5 g/dL for males
    2. White blood cells (WBC) range: 3,500-9,000 cells/mm^3
    3. Platelets between 150,000 - 450,000 cells/µL
    4. Normal liver function: Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤1.25x upper limit of normal
    5. Serum creatinine ≤1.25x upper limit of normal
    6. Urinalysis: blood and protein less than 1+ and negative glucose
    7. Negative HIV serology Note: HIV serology testing will be done via enzyme immunoassay with confirmatory testing of reactive results through a repeat enzyme immunoassay followed by an antibody differentiation immunoassay. After the repeat enzyme immunoassay, if an antibody differentiation immunoassay cannot be done for any reason, then confirmatory testing will be done via Western Blot. HIV rapid testing will not be performed in this study.
    8. Negative hepatitis B surface antigen (HbsAg)
    9. Negative hepatitis C serology or negative hepatitis C RNA (viral load) if antibodies are detected Note: Each laboratory screening test that is out of acceptable range can be repeated one time during the screening window if there is a possible alternative explanation for the out of range value or if the out of range value is due to a temporary condition that resolves within the screening visit window. A second screening visit may be conducted outside of the initial screening visit window for volunteers who meet certain criteria if study enrollment and/or participant replacement is ongoing.
11. Biological Male-Specific Criteria:

    1. Must agree to refrain from donating sperm from screening until at least 12 weeks after the last study injection
    2. Must agree to consistently use a method of contraception from screening until at least 12 weeks after the last study injection
12. Biological Female-Specific Criteria:

    1. Not pregnant within 12 weeks prior to screening, not pregnant or breastfeeding at screening, and not planning to become pregnant or breastfeed at any time from screening until 12 weeks after the last study injection
    2. Must have a negative human chorionic gonadotropin (β-HCG) pregnancy test (urine) at screening and at timepoints throughout the study, if of childbearing potential
    3. Must agree to consistently practice a highly effective method of contraception at least 45 days prior to enrollment and for 12 weeks after the final injection, if of childbearing potential

Exclusion Criteria:

Volunteers will be excluded if any of the following apply:

1. Body mass index (BMI) <18.0 kg/m^2 and >35.1 kg/m^2
2. Has a condition which affects immune function, including but not limited to:

   1. Known or suspected congenital or acquired immunodeficiency
   2. Diabetes mellitus type 1 or type 2 (including cases controlled with diet alone) Note: A history of isolated gestational diabetes is not an exclusion criterion.
   3. Thyroid disease
   4. Asplenia, defined as any condition resulting in the absence of a functional spleen
   5. Conditions and diagnoses defined as potential immune-mediated medical conditions
3. Has a history of other chronic or clinically significant diseases or medical conditions that in the opinion of the investigator would jeopardize the safety or rights of the participant Note: Includes but is not limited to sickle cell anemia, chronic hepatitis or cirrhosis, chronic urticaria, chronic cardiac disease, hypertension not controlled by medication, severe asthma, chronic pulmonary disease, renal failure, and lymphatic filariasis.
4. Has a history of malignancy other than squamous cell or basal cell skin cancer, unless there has been definitive surgical and/or medical treatment that is considered to have achieved a cure
5. Had major surgery (per the physician investigator's judgment) within the 28 days prior to screening or has plans to have major surgery during the study
6. Has a personal or family history of a bleeding disorder, such as factor deficiency, coagulopathy, or platelet disorder requiring special precautions
7. Has a personal or family history of a blood clotting disorder, such as thrombosis with thrombocytopenia syndrome (TTS), heparin-induced thrombocytopenia and thrombosis (HITT), deep vein thrombosis, pulmonary embolism, acute myocardial infarction, and stroke
8. Has a condition known to increase risk of blood clotting, including but not limited to autoimmune disease, connective tissue and other inflammatory conditions, immobility, recent infection, and recent head trauma including cerebrovascular accidents (stroke)
9. Hepatitis B surface antigen positive at any time in the past
10. Untreated syphilis infection as confirmed by RPR or a similar quantitative nontreponemal test such as VDRL
11. Prior receipt or plans to receive any of the following:

    1. Chronic use of therapies that may modify immune response, such as high dose inhaled and sprayed corticosteroids (>440 µg/twice daily doses of inhaled fluticasone equivalent) and systemic corticosteroids (>20 mg/day doses of prednisone equivalent for periods exceeding 10 days) within 14 days prior to enrollment or at any time during participation in this study Note: The following exceptions are permitted and will not exclude study participation: use of stable low/medium doses (<440 µg/twice daily doses of inhaled fluticasone equivalent) of inhaled and sprayed corticosteroids, topical corticosteroids for an acute uncomplicated dermatitis; or a short course (duration of 10 days or less, or a single injection) of corticosteroid for a non-chronic condition (based on the physician investigator's clinical judgment) at least 14 days prior to enrollment in this study. Includes other medications, which, in the opinion of the physician investigator(s), will impact the participant's immune response.
    2. Blood products within 120 days prior to enrollment or at any time during participation in this study
    3. Immunoglobulins within 90 days prior to enrollment or at any time during participation in this study
    4. Therapy for active tuberculosis within 90 days prior to enrollment, unless the therapy is considered to have achieved a cure, or at any time during participation in this study
    5. Licensed or authorized vaccine from 30 days prior to enrollment until 42 days (6 weeks) after the last study injection Note: Participants may receive inactivated seasonal influenza vaccine or COVID-19 vaccine during their participation in this study but not within 14 days prior or 6 weeks after each study injection
    6. Any investigational study products for conditions other than HIV within 90 days prior to enrollment or at any time during participation in this study
    7. An investigational HIV vaccine or HIV antibody at any time prior to or during participation in this study
    8. Medications that increase the risk of bleeding (warfarin, clopidogrel, ticagrelor, dabigatran, rivaroxaban, apixaban, heparin and other heparinoids) or blood clots (heparin in participants who have a prior history of heparin-induced coagulopathy) within 30 days prior to enrollment or at any time during participation in this study. [Note: Volunteers determined to be ineligible at screening due to receipt of the above listed substances may be re-screened once the applicable window of receipt has expired if study enrollment and/or participant replacement is ongoing].
12. Has a known allergy or history of anaphylaxis or other serious reaction to a vaccine, vaccine component, or latex
13. Current or planned participation in another study requiring blood draws or exposure to investigational or non-investigational vaccine/product (pharmaceutical or device) throughout the study period
14. Has tattoos, scars, or other marks that would, in the opinion of the physician investigator, interfere with the assessment of the injection sites
15. Current or history of substance abuse within 12 months prior to enrollment that, in the physician investigator's opinion, could interfere with reliable participation
16. In the physician investigator's opinion, is unable to communicate reliably, is unlikely to adhere to study requirements, or has a condition that would limit completion of the study
17. Any other chronic or clinically significant medical condition that in the opinion of investigator would jeopardize the safety or rights of the participant or potentially impairs immune response or threatens conduct of the study according to protocol
18. Study site employee

Final evaluation of eligibility will be based on the medical judgment of the physician investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence and severity of solicited local and systemic adverse events (AEs) following candidate vaccine administration | Day 0 - Day 505
  Occurrence and severity of solicited local and systemic adverse events (AEs) following candidate vaccine administration.
Occurrence, severity, and relationship to vaccination of unsolicited adverse events after candidate vaccine administration | Day 0 - Day 505
  Occurrence, severity, and relationship to vaccination of unsolicited adverse events after candidate vaccine administration.
Occurrence of serious adverse events (SAEs) following candidate vaccine administration | Day 0 - Day 505
  Occurrence of serious adverse events (SAEs) following candidate vaccine administration.
Occurrence of adverse events of special interest (AESIs) following candidate vaccine administration | Day 0 - Day 505
  Occurrence of adverse events of special interest (AESIs) following candidate vaccine administration.

SECONDARY OUTCOMES:
Quantify IgG binding antibodies to HIV Env in terms of magnitude, breadth, and durability between Arms | Visit Days 1, 4, 8, 15, 29, 57, 71, 85,169, 183, and 337
  Quantify IgG binding antibodies to HIV Env in terms of magnitude between Arms. HIV-specific Binding Antibody ELISA Assays will be performed to detect plasma IgG and IgA binding antibodies to HIV-1 Envelope antigens and assess their magnitude between Arms.
Quantify neutralizing antibodies to HIV Env in terms of magnitude, breadth, and durability between Arms | Visit Days 1, 4, 8, 15, 29, 57, 71, 85,169, 183, and 337
  Quantify rate of neutralizing antibodies to HIV Env in terms of magnitude between Arms. Neutralizing Antibody Assays will be measured as a function of reductions in luciferase (Luc) reporter gene expression after a single round of infection in TZM-bl cells using high throughput analysis.

OTHER OUTCOMES:
Characterize binding antibody Fc engagement to a panel of HIV Envs as assessed by Antibody Profiling | Visit Days 1, 15, 29, 57, 71, 85, 169, 183, and 337
  Characterize binding antibody Fc engagement to a panel of HIV Envs. Antibody Profiling will be conducted to assess antibody breadth and correlation of Fc receptor usage with antibody function.The current capacity for Antibody Profiling is the assessment of over 300 samples in one experiment. The beads presenting the HIV antigens will be distributed robotically in a high-throughput manner into 384 well plates. Similarly, the samples will be diluted robotically and incubated with the beads. Detection reagents will be added to the wells after washing. These detection reagents are inclusive of subclass, isotype, and Fc receptor usage.
Characterize rate of B-cell specificity by quantifying antigen-specific responses as assessed through B-cell ELISPOT | Visit Days 1, 8, 15, 29, 71, 169, 176, 183, and 337
  Characterize rate of B-cell specificity by quantifying antigen-specific responses as assessed through B-cell ELISPOT
Characterize magnitude of cell-mediated immune responses elicited across vaccination regimens (including antigen -specific CD4 and CD8 T cell responses) assessed by CD4 and CD8 cellular response assays and after stimulation with HIV-specific antigens. | Visit Days 1, 4, 8, 29, 71, 169, 170, 176, 183, and 337
  Characterize and assess the magnitude of cell-mediated immune responses elicited across vaccination regimens including but not limited to antigen -specific CD4 and CD8 T cell responses as assessed by CD4 and CD8 cellular response assays and after stimulation with HIV-specific antigens.
Phenotype innate immune cells (NK cells) as assessed by flow cytometry | Visit Days 1, 4, 8, 29, 71, 169, 170, 176, 183, and 337
  Characterize cytokines elicited by vaccine regimens

CONTACTS AND LOCATIONS:
Overall Officials: Grace Mirembe, MBChB, MMed, Principal Investigator — Makerere University Walter Reed Project P.O. Box 16524, Kampala, Uganda
Locations (1):
- Makerere University Walter Reed Project (MUWRP), Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pitisuttithum P, Gilbert P, Gurwith M, Heyward W, Martin M, van Griensven F, Hu D, Tappero JW, Choopanya K; Bangkok Vaccine Evaluation Group. Randomized, double-blind, placebo-controlled efficacy trial of a bivalent recombinant glycoprotein 120 HIV-1 vaccine among injection drug users in Bangkok, Thailand. J Infect Dis. 2006 Dec 15;194(12):1661-71. doi: 10.1086/508748. Epub 2006 Nov 3. PMID 17109337
- [Background] Pauthner M, Havenar-Daughton C, Sok D, Nkolola JP, Bastidas R, Boopathy AV, Carnathan DG, Chandrashekar A, Cirelli KM, Cottrell CA, Eroshkin AM, Guenaga J, Kaushik K, Kulp DW, Liu J, McCoy LE, Oom AL, Ozorowski G, Post KW, Sharma SK, Steichen JM, de Taeye SW, Tokatlian T, Torrents de la Pena A, Butera ST, LaBranche CC, Montefiori DC, Silvestri G, Wilson IA, Irvine DJ, Sanders RW, Schief WR, Ward AB, Wyatt RT, Barouch DH, Crotty S, Burton DR. Elicitation of Robust Tier 2 Neutralizing Antibody Responses in Nonhuman Primates by HIV Envelope Trimer Immunization Using Optimized Approaches. Immunity. 2017 Jun 20;46(6):1073-1088.e6. doi: 10.1016/j.immuni.2017.05.007. PMID 28636956
- [Background] Liao HX, Lynch R, Zhou T, Gao F, Alam SM, Boyd SD, Fire AZ, Roskin KM, Schramm CA, Zhang Z, Zhu J, Shapiro L; NISC Comparative Sequencing Program; Mullikin JC, Gnanakaran S, Hraber P, Wiehe K, Kelsoe G, Yang G, Xia SM, Montefiori DC, Parks R, Lloyd KE, Scearce RM, Soderberg KA, Cohen M, Kamanga G, Louder MK, Tran LM, Chen Y, Cai F, Chen S, Moquin S, Du X, Joyce MG, Srivatsan S, Zhang B, Zheng A, Shaw GM, Hahn BH, Kepler TB, Korber BT, Kwong PD, Mascola JR, Haynes BF. Co-evolution of a broadly neutralizing HIV-1 antibody and founder virus. Nature. 2013 Apr 25;496(7446):469-76. doi: 10.1038/nature12053. Epub 2013 Apr 3. PMID 23552890
- [Background] Havenar-Daughton C, Carnathan DG, Torrents de la Pena A, Pauthner M, Briney B, Reiss SM, Wood JS, Kaushik K, van Gils MJ, Rosales SL, van der Woude P, Locci M, Le KM, de Taeye SW, Sok D, Mohammed AUR, Huang J, Gumber S, Garcia A, Kasturi SP, Pulendran B, Moore JP, Ahmed R, Seumois G, Burton DR, Sanders RW, Silvestri G, Crotty S. Direct Probing of Germinal Center Responses Reveals Immunological Features and Bottlenecks for Neutralizing Antibody Responses to HIV Env Trimer. Cell Rep. 2016 Nov 22;17(9):2195-2209. doi: 10.1016/j.celrep.2016.10.085. PMID 27880897
- [Background] Genito CJ, Beck Z, Phares TW, Kalle F, Limbach KJ, Stefaniak ME, Patterson NB, Bergmann-Leitner ES, Waters NC, Matyas GR, Alving CR, Dutta S. Liposomes containing monophosphoryl lipid A and QS-21 serve as an effective adjuvant for soluble circumsporozoite protein malaria vaccine FMP013. Vaccine. 2017 Jul 5;35(31):3865-3874. doi: 10.1016/j.vaccine.2017.05.070. Epub 2017 Jun 7. PMID 28596090
- [Background] Cirelli KM, Carnathan DG, Nogal B, Martin JT, Rodriguez OL, Upadhyay AA, Enemuo CA, Gebru EH, Choe Y, Viviano F, Nakao C, Pauthner MG, Reiss S, Cottrell CA, Smith ML, Bastidas R, Gibson W, Wolabaugh AN, Melo MB, Cossette B, Kumar V, Patel NB, Tokatlian T, Menis S, Kulp DW, Burton DR, Murrell B, Schief WR, Bosinger SE, Ward AB, Watson CT, Silvestri G, Irvine DJ, Crotty S. Slow Delivery Immunization Enhances HIV Neutralizing Antibody and Germinal Center Responses via Modulation of Immunodominance. Cell. 2019 May 16;177(5):1153-1171.e28. doi: 10.1016/j.cell.2019.04.012. Epub 2019 May 9. PMID 31080066

DOCUMENTS (4):
  • Informed Consent Form: Future Use ICF V1.4 dated 12JUL24 (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT06205056/ICF_000.pdf
  • Informed Consent Form: Optional Lymph Node Biopsy ICF V1.4 dated 12JUL24 (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT06205056/ICF_001.pdf
  • Informed Consent Form: Genetic ICF V1.4 dated 12JUL24 (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT06205056/ICF_002.pdf
  • Informed Consent Form: Main ICF V1.4 dated 12JUL24 (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT06205056/ICF_003.pdf